CLINICAL TRIAL: NCT05567653
Title: Effects of 3-month Probiotic Mix Supplementation (L. Helveticus R-0052, B. Longum R-0175) on Gut Microbiota and Metabolome, Endocannabinoid and Immune Systems Activation, Along With Symptoms of Fatigue in Professional Dancers
Brief Title: Effects of Probiotics on Gut Microbiota, Endocannabinoid and Immune Activation and Symptoms of Fatigue in Dancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Jakub Wiącek, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11/NSN/4/2022
Record Dates: First submitted 2022-09-22; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Fatigue; Stress, Job
Keywords: Gut microbiome; Probiotics; Professional dancers; Cannabinoids; Inflammation
MeSH Terms: conditions — Fatigue; Occupational Stress; Inflammation | interventions — Starch

STUDY DESIGN:
Intervention Model Description: a Randomized, Double-blind, Placebo-controlled Study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic treatment group (Experimental): ca. 30 participants
  Interventions: Dietary Supplement: Lactobacillus helveticus Rosell-52 and Bifidobacterium longum Rosell-175 (Sanprobi Stress)
- Placebo group (Placebo Comparator): ca. 30 participants
  Interventions: Dietary Supplement: Starch (placebo)

INTERVENTIONS:
Dietary Supplement: Lactobacillus helveticus Rosell-52 and Bifidobacterium longum Rosell-175 (Sanprobi Stress) — 3-month, multi-strain probiotic supplementation (one a day, 3 x 10⁹ CFU)
  Other Names: L. helveticus R-0052, B. longum R-0175
  Arms: Probiotic treatment group
Dietary Supplement: Starch (placebo) — 3-month placebo
  Other Names: capsules containing starch
  Arms: Placebo group

SUMMARY:
The aim of the planned research is to assess the dynamics of changes in the elements of the gut-brain axis (GBA), the cytokine profile and the endocannabinoid system markers, after dietary supplementation with probiotics Lactobacillus helveticus Rosell-52 and Bifidobacterium longum Rosell-175 by professional dancers. Although in recent years there has been growing interest in the influence of the gut microbiota on the body's adaptation to stress stimuli and on overall health, there is a lack of information on the influence of probiotics on systems involved in maintaining neuropsychiatric balance, such as the endocannabinoid system.

In order to determine the validity of the applied therapy with selective probiotics, the following will be assessed: intestinal bacteria and bacterial metabolites in the stool, cannabinoids and cannabinoid receptors and enzymes in the blood, indicators of mental distress in the blood, cytokines responsible for the modulation of the gut-brain axis in the blood, as well as questionnaires regarding the functioning of the digestive tract, fatigue, stress and sleep quality.

The study will involve active dancers of the Polish Theater in Poznan, the Polish Dance Theater, the Private School of Dance Art in Poznan and students of the Academy of Physical Education in the field of Dance. Dancers are a group of athletes that is exposed to particular injuries and work-overload. Professional dancers spend multiple hours a week on intensive physical training. The largest percentage of injuries occurring in the group of professional dancers are chronic injuries, including: inflammation of soft tissues, muscle strains and tears.

Professional dance is one of the most physically demanding forms of physical activity, and at the same time it is associated with a high burden on the nervous system problems caused by performances in front of an audience or subjective jury, frequent traveling and disturbances in the circadian rhythm.

DETAILED DESCRIPTION:
Professional dancers are often referred to as artistic athletes due to their high level of physical activity and competition. Training dance for over 11.5 hours a week increases the risk of injury (women - mostly bone injuries, men - mostly bruises and tendon injuries). One of the reasons for the increased susceptibility to injuries among dancers is psychological stress. The observations results indicate that dancers often decide to continue training despite feeling pain, which limits the smoothness of their movements and leads to a further increase of stress. Highly physically active groups of people are more exposed to functional dyspepsia (FD) and irritable bowel syndrome (IBS), which occurence is correlated to chronic stress. As a result of chronic stress and the activation of the hypothalamic pituitary-adrenal axis (HPA), inflammatory processes in the gastrointestinal mucosa are initiated. The presence of noradrenaline increases the adhesion of bacteria and viruses to the epithelium, which in turn modulates the immune system within the intestines and increases their inflammation. Systemically acting cortisol causes the leakage of tight junctions (TJ) cells and an increase in the permeability of the intestinal barrier. Inflammation stimulates the secretion of cortisol, which initiates the further cycle of inflammation and weakening of the intestinal barrier function. As a consequence, cytokines and inflammatory mediators released in the course of inflammation act directly on the nerve endings that transmit these afferent nerve signals to the brain, becoming an endogenous stressor.

When exogenous and endogenous stress factors overlap, the body's perception of stress increases, which ultimately leads to psychological, physiological and behavioral changes.

Pain and depression are common comorbidities of neuropsychiatric origin. One of the body's regulatory systems, which in both cases is dysfunctional, is the endocannabinoid system (ECS). It has been suggested that these diseases can be caused by intense and prolonged exercise, which disrupts the intestinal barrier, causing changes in the profile of metabolites and the function of the intestinal microbiota. Overtraining leads to an increase in the levels of cortisol, adrenaline and noradrenaline, and to the translocation of lipopolysaccharide (LPS) outside the gut, increasing the concentration of pro-inflammatory cytokines in the body. This results in dysregulation of the balance between serotonin (5-HT), dopamine (DA) and gamma-aminobutyric acid (GABA) and fatigue. These changes lead to further activation of the endocannabinoid system and, in the long-term, weakening of adaptive abilities.

The neuromodulatory properties of the cannabinoid system are manifested e.g. in short- and long-term synaptic plasticity and modulation of pain conduction. Research results indicate that the endocannabinoid system, in addition to its key role in regulating intestinal motility, also affects the secretory functions of the gastrointestinal tract and the integrity of the intestinal epithelium, which may be an alternative way to regulate the immune system and inflammation in the intestines.

Type 1 cannabinoid receptors (CB1) are located presynaptically in the cell membrane of central and peripheral nervous system neurons, and their activation inhibits the release of many neurotransmitters, i.e. acetylcholine, noradrenaline, dopamine, serotonin, glutamate and γ-aminobutyric acid. Type 2 cannabinoid receptors (CB2) are found mainly on the surface of cells of the immune system, especially B-lymphocytes, macrophages and monocytes. Their activation inhibits pro-inflammatory cytokines release and increases the release of anti-inflammatory cytokines.

Cannabinoid receptors are found in both, the immune and digestive systems. Endogenous cannabinoids modify the body's response to stress by influencing the hypothalamic pituitary-adrenal axis (HPA). Stress leads to an increased activity of endocannabinoids which, mainly through the CB1 cannabinoid receptors, lead to the inhibition of the release of corticosteroids. In addition, the activation of CB1 receptors in the gastrointestinal tract reduces the intensity of pain conduction (nociception), which is induced by activation, e.g. TRPV1 vanilloid receptors. It has been shown that inflammation within the intestinal epithelium of the gastrointestinal tract causes an increase in the neural conduction of neurons containing CB1 receptors, which contributes to a change in the proportion of these receptors in relation to the TRPV1 located mainly in the cell membrane of dorsal root ganglion afferents (DRGs). As a result, two different receptors interact and the TRPV1 receptor activity is abolished. Inflammatory mediators released from the intestinal epithelium stimulate visceral pain, while activation of CB2 receptors probably reduces their action.

There are indications that a qualitative and quantitative change in the intestinal microbiota may affect the activity of endogenous ligands and mediators of the endocannabinoid system (ECS). Although the mechanisms of regulation of the level of endocannabinoids and related bioactive lipids by selected bacteria are not fully understood, it has been shown that probiotic supplementation can induce an increase in the concentration of endogenous cannabinoids, i.e. 2-AG, 2-OG (oleoylglycerol) and 2-PG (palmitoylglycerol). In an animal experiment, the use of monoacylglycerol lipase inhibition reduced the degradation of 2-AG, which reduced endotoxemia and systemic inflammation. In another study, the deletion of the Myd88 gene encoding the TLR (toll-like receptor) receptor protein in intestinal epithelial cells changed the composition of the intestinal microbiota, decreased the synthesis of anandamide (AEA) and increased the synthesis of anti-inflammatory endocannabinoids, such as: 2-AG, 2-PG, 2 OG. Released endocannabinoids with anti-inflammatory properties have the ability to activate so-called orphan GPR119 receptors, which are associated with the secretion of anti-inflammatory mediators. Moreover, it has been shown that an increase in LPS concentration induces AEA synthesis and a decrease in fatty-acid amide hydrolase (FAAH) in macrophages, as well as an increase in AEA production in peripheral lymphocytes, which may be important for the regulation of the intestinal barrier function and the level of inflammation. The results of studies carried out on a mouse model revealed the importance of the intestinal microbiota in the regulation of the expression of the NAPE-PLD gene (phospholipase D specific for n-acylphosphatidylethanolamine), i.e. an enzyme involved in the synthesis of anandamide and in the selective regulation of CB1 mRNA expression. In an obese mouse model, it was observed that the administration of a probiotic decreased the expression level of CB1 receptor mRNA while reducing the concentration of AEA ligand and increasing the expression of FAAH mRNA. In other studies, administration of a probiotic to mice resulted in a decrease in the concentration of LPS in the blood plasma, which correlated with both the level of AEA and the expression of CB1 mRNA in the colon epithelium. In in vitro and in vivo experiments on animal models, it has been observed that CB2 receptors are activated when an imbalance in the innate immune system occurs. The NLRP3 inflammasomes are suppressed by autophagy, a mechanism that may be involved in the suppression of inflammation and the regulation of the intestinal barrier, e.g. in irritable bowel syndrome. Another factor that is a potential NLRP3 inhibitor is the intestinal microbiota metabolite, butyrate, which belongs to the short-chain fatty acids. Its action has a positive effect on the functions of the intestinal epithelial cells and the stability of the intestinal barrier. In studies conducted on germ-free mice, after the intestinal microbiota was transferred, the metabolism of endocannabinoids in the gastrointestinal tract changed. The use of probiotic therapy in mice with previously induced intestinal dysbiosis changed the activation of endocannabinoid receptors, the behavior of animals and a decrease in intestinal inflammation. Other research results indicate that inhibition of the CB1 receptor in obese mice stimulates the secretion of mucin, which is the primary source of nutrients for the development of Akkermansia muciniphila. This observation confirms the results of studies by other authors, who demonstrated the possibility of regulation of CB2 receptors by some species of intestinal bacteria and the related immune response.

The mechanisms of the transmission of inflammatory signals from the gut to the CNS are not fully elucidated. The results of the research indicate, however, that the systemic inflammation accompanying depressive symptoms is associated with changes in the ecosystem of the intestinal microbiota and the production of SCFA and other metabolites of a neurobiological nature. Moreover, it can also lead to changes in the synthesis and release of endocannabinoids or the metabolic pathways of tryptophan and kynurenine (KYN). So far, it has been observed that there is a link between ECS and the kynurenine pathway in neurological disorders such as epilepsy or migraine headaches, which are associated with excessive cell stimulation and excitotoxicity. The latest research results indicate the possibility of modifying the transformations of tryptophan and kynurenine by probiotic therapy.

There is limited number of human research on the role of the gut microbiota in the modulation of the ECS. The available literature lacks studies describing the relationship of changes in the intestinal microbiota and its metabolome under the influence of targeted, multi-strain probiotic therapy on the response of the endocannabinoid and immune system in people subjected to high physical and mental stress. Observations that will be made in dancers supplemented with a multi strain probiotic containing Lactobacillus helveticus Rosell-52 and Bifidobacterium longum Rosell-175 may help finding effective tools in the treatment of gastrointestinal disorders and stress related to it. A potential mechanism behind this action may be the restoration of the normal gut microbiota and the profile of its metabolites, as well as the improvement of the gut barrier and endocannabinoid function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, <36 years old;
* Professional dancing activity with over 8 hours of training per week.

Exclusion Criteria:

* Age <18,> 36 y.o.;
* Being injured within 3 months from the start of the study;
* Taking pre- and / or probiotics in the last 3 months before the study;
* Hospitalization during the last 4 weeks before starting of the study;
* Traveling to tropical countries during the last 4 weeks before study;
* Taking antibiotics, steroids and anabolic steroids in the last 4 weeks before study.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of intestinal microbiota in stool samples | up to 10 months
  • gut bacteria species in stool will be assessed using the shallow shotgun sequencing method, NGS (Next Generation Sequencing);
Quantitive change in intestinal microbiota in stool samples | up to 10 months
  • determination of quantitative (Colony forming units - CFU) changes in bacteria in the stool - the shallow shotgun sequencing method, NGS (Next Generation Sequencing) molecular analysis will be used to assess the changes;
Intestinal metabolome in stool samples | up to 10 months
  • metabolomic analysis (non-targeted metabolome, short-chain fatty acids, trimethylamines, tryptophan catabolites) will be performed on a quadrupole mass spectrometer coupled with a time-of-flight (QToF) analyzer connected to the AB Sciex - TripleTOF® 6600+ high performance liquid chromatograph (UHPLC)
Quantitive change in endocannabinoids levels in blood samples | up to 10 months
  • determination of endocannabinoids and cannabinoid receptors: anandamide (AEA) and 2-arachidonylglycerol (2-AG) using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in endocannabinoids' receptors levels in blood samples | up to 10 months
  • determination of cannabinoid receptors: Endocannabinoid Receptor 1 (CNR1) and Endocannabinoid Receptor 2 (CNR2) using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in endocannabinoids metabolism enzymes in blood | up to 10 months
  • determination of cannabinoid metabolism enzymes: fatty acid amide hydrolase (FAAH) and monoacylglycerol lipase (MAGL) using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in intestinal barrier proteins in blood samples | up to 10 months
  • determination of blood biomarkers of a disturbed intestinal barrier concentrations: zonulin, calprotectin (CALPRO) using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in intestinal barrier biomarkers in blood samples | up to 10 months
  • determination of blood biomarkers of a disturbed intestinal barrier concentrations: lipopolysaccharide (LPS), secretory immunoglobulin A (sIgA) using ELISA Kit (picograms per millilitre (pg/mL));
Quantitive change in tumor necrosis factor-alpha (TNF-α) in blood samples | up to 10 months
  • determination of blood tumor necrosis factor-alpha (TNF-α) concentration using leukemia inhibitory factor (LIF) concentration using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in leukemia inhibitory factor (LIF) in blood samples | up to 10 months
  • determination of blood leukemia inhibitory factor (LIF) concentration using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in blood interleukins profile | up to 10 months
  • determination of interleukins concentrations: IL-1α, IL-1β, IL-10 and IL-18 using ELISA Kit using ELISA Kit (picograms per millilitre (pg/mL));
Quantitive change in chronic stress biomarker in blood samples - cortisol | up to 10 months
  • determination of blood cortisol concentration using ELISA Kit (nanograms per millilitre (ng/mL));
Quantitive change in inflammation biomarker in blood samples - C-reactive protein | up to 10 months
  • determination of C-reactive protein (CRP) concentration using ELISA Kit (picograms per millilitre (pg/mL));

SECONDARY OUTCOMES:
Coping with stress questionnaire | up to 10 months
  • determination of methods of coping with stress using the Inventory for Measuring Coping with Stress (Mini-COPE); It is designed to establish how a study participant behaves when experiences particular events; The scale: 0 = "I hardly ever do this", 1 = "I rarely do this", 2 = "I do this often", 3 = "I almost always do this";
Fatigue questionnaire | up to 10 months
  • assessment of the level of fatigue using the Fatigue Assessment Scale (FAS); the statements of the questionnaire relate to the feeling of well-being; The scale: 1. Never, 2. Sometimes (once a month or less), 3. Regularly (several times a month), 4. Often (weekly) and 5. Always (everyday);
Gastrointestinal disorders questionnaire | up to 10 months
  • assessment of gastrointestinal disorders using the Rome IV Questionnaire for adults (selected questions on irritable bowel syndrome, constipation and diarrhea); the statements of the questionnaire relate to frequency and intensity of disorders; higher scores mean worse outcome;
Sleep quality questionnaire | up to 10 months
  • assessment of the sleep quality level using Pittsburgh Sleep Quality Questionnaire, PSQI; the statements of the questionnaire relate to frequency of sleep disorders; higher scores mean worse outcome;
Body mass analysis (BMI, kg/m^2) | up to 10 months
  • determination of body weight and composition using the electrical bioimpedance method;
Body composition analysis (percent of total body mass) | up to 10 months
  • assessment of bone, fat and fat-free mass using the electrical bioimpedance method;
Composite measure of Diet composition assessed by food diaries | up to 10 months
  • assessment of protein, fat, carbohydrates and fibre intake using food diaries (grams);
Pain threshold test (Newtons) | up to 10 months
  • mechanical stimuli pain threshold assessment using an algometer (Wagner FPX ™)
Changes in red blood cells count | up to 10 months
  • determination of red blood cell counts using flow cytometry (trillion cells per Litre);
Changes in white blood cells count | up to 10 months
  • determination of white blood cells counts using flow cytometry (billion cells per Litre);
Changes in hemoglobin level | up to 10 months
  • determination of hemoglobin level using flow cytometry (grams per Litre);
Changes in hematocrit | up to 10 months
  • determination of hematocrit using flow cytometry (percentage of red blood cells in blood);
Changes in platelets counts | up to 10 months
  • determination of platelets counts using flow cytometry (billions per Litre)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Karolkiewicz, Professor, Study Chair — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acharya N, Penukonda S, Shcheglova T, Hagymasi AT, Basu S, Srivastava PK. Endocannabinoid system acts as a regulator of immune homeostasis in the gut. Proc Natl Acad Sci U S A. 2017 May 9;114(19):5005-5010. doi: 10.1073/pnas.1612177114. Epub 2017 Apr 24. PMID 28439004
- [Background] Alhouayek M, Muccioli GG. COX-2-derived endocannabinoid metabolites as novel inflammatory mediators. Trends Pharmacol Sci. 2014 Jun;35(6):284-92. doi: 10.1016/j.tips.2014.03.001. Epub 2014 Mar 29. PMID 24684963
- [Background] Alhouayek M, Lambert DM, Delzenne NM, Cani PD, Muccioli GG. Increasing endogenous 2-arachidonoylglycerol levels counteracts colitis and related systemic inflammation. FASEB J. 2011 Aug;25(8):2711-21. doi: 10.1096/fj.10-176602. Epub 2011 May 6. PMID 21551239
- [Background] Biernacki M, Skrzydlewska E. Metabolism of endocannabinoids. Postepy Hig Med Dosw (Online). 2016 Aug 11;70(0):830-43. doi: 10.5604/17322693.1213898. PMID 27516570
- [Background] Cani PD, Plovier H, Van Hul M, Geurts L, Delzenne NM, Druart C, Everard A. Endocannabinoids--at the crossroads between the gut microbiota and host metabolism. Nat Rev Endocrinol. 2016 Mar;12(3):133-43. doi: 10.1038/nrendo.2015.211. Epub 2015 Dec 18. PMID 26678807
- [Background] Cani PD, Bibiloni R, Knauf C, Waget A, Neyrinck AM, Delzenne NM, Burcelin R. Changes in gut microbiota control metabolic endotoxemia-induced inflammation in high-fat diet-induced obesity and diabetes in mice. Diabetes. 2008 Jun;57(6):1470-81. doi: 10.2337/db07-1403. Epub 2008 Feb 27. PMID 18305141
- [Background] Cani PD, Possemiers S, Van de Wiele T, Guiot Y, Everard A, Rottier O, Geurts L, Naslain D, Neyrinck A, Lambert DM, Muccioli GG, Delzenne NM. Changes in gut microbiota control inflammation in obese mice through a mechanism involving GLP-2-driven improvement of gut permeability. Gut. 2009 Aug;58(8):1091-103. doi: 10.1136/gut.2008.165886. Epub 2009 Feb 24. PMID 19240062
- [Background] Castillo PE, Younts TJ, Chavez AE, Hashimotodani Y. Endocannabinoid signaling and synaptic function. Neuron. 2012 Oct 4;76(1):70-81. doi: 10.1016/j.neuron.2012.09.020. PMID 23040807
- [Background] Caporaso JG, Kuczynski J, Stombaugh J, Bittinger K, Bushman FD, Costello EK, Fierer N, Pena AG, Goodrich JK, Gordon JI, Huttley GA, Kelley ST, Knights D, Koenig JE, Ley RE, Lozupone CA, McDonald D, Muegge BD, Pirrung M, Reeder J, Sevinsky JR, Turnbaugh PJ, Walters WA, Widmann J, Yatsunenko T, Zaneveld J, Knight R. QIIME allows analysis of high-throughput community sequencing data. Nat Methods. 2010 May;7(5):335-6. doi: 10.1038/nmeth.f.303. Epub 2010 Apr 11. No abstract available. PMID 20383131
- [Background] Cheng YH, Ho MS, Huang WT, Chou YT, King K. Modulation of Glucagon-like Peptide-1 (GLP-1) Potency by Endocannabinoid-like Lipids Represents a Novel Mode of Regulating GLP-1 Receptor Signaling. J Biol Chem. 2015 Jun 5;290(23):14302-13. doi: 10.1074/jbc.M115.655662. Epub 2015 Apr 22. PMID 25903129
- [Background] Colin-Gonzalez AL, Aguilera G, Santamaria A. Cannabinoids: Glutamatergic Transmission and Kynurenines. Adv Neurobiol. 2016;12:173-98. doi: 10.1007/978-3-319-28383-8_10. PMID 27651254
- [Background] Crowe MS, Nass SR, Gabella KM, Kinsey SG. The endocannabinoid system modulates stress, emotionality, and inflammation. Brain Behav Immun. 2014 Nov;42:1-5. doi: 10.1016/j.bbi.2014.06.007. Epub 2014 Jun 19. PMID 24953427
- [Background] Derrien M, Vaughan EE, Plugge CM, de Vos WM. Akkermansia muciniphila gen. nov., sp. nov., a human intestinal mucin-degrading bacterium. Int J Syst Evol Microbiol. 2004 Sep;54(Pt 5):1469-1476. doi: 10.1099/ijs.0.02873-0. PMID 15388697
- [Background] Everard A, Belzer C, Geurts L, Ouwerkerk JP, Druart C, Bindels LB, Guiot Y, Derrien M, Muccioli GG, Delzenne NM, de Vos WM, Cani PD. Cross-talk between Akkermansia muciniphila and intestinal epithelium controls diet-induced obesity. Proc Natl Acad Sci U S A. 2013 May 28;110(22):9066-71. doi: 10.1073/pnas.1219451110. Epub 2013 May 13. PMID 23671105
- [Background] Everard A, Geurts L, Caesar R, Van Hul M, Matamoros S, Duparc T, Denis RG, Cochez P, Pierard F, Castel J, Bindels LB, Plovier H, Robine S, Muccioli GG, Renauld JC, Dumoutier L, Delzenne NM, Luquet S, Backhed F, Cani PD. Intestinal epithelial MyD88 is a sensor switching host metabolism towards obesity according to nutritional status. Nat Commun. 2014 Dec 5;5:5648. doi: 10.1038/ncomms6648. PMID 25476696
- [Background] Fitzgibbon M, Finn DP, Roche M. High Times for Painful Blues: The Endocannabinoid System in Pain-Depression Comorbidity. Int J Neuropsychopharmacol. 2015 Sep 5;19(3):pyv095. doi: 10.1093/ijnp/pyv095. PMID 26342110
- [Background] Forteza F, Giorgini G, Raymond F. Neurobiological Processes Induced by Aerobic Exercise through the Endocannabinoidome. Cells. 2021 Apr 17;10(4):938. doi: 10.3390/cells10040938. PMID 33920695
- [Background] Guida F, Turco F, Iannotta M, De Gregorio D, Palumbo I, Sarnelli G, Furiano A, Napolitano F, Boccella S, Luongo L, Mazzitelli M, Usiello A, De Filippis F, Iannotti FA, Piscitelli F, Ercolini D, de Novellis V, Di Marzo V, Cuomo R, Maione S. Antibiotic-induced microbiota perturbation causes gut endocannabinoidome changes, hippocampal neuroglial reorganization and depression in mice. Brain Behav Immun. 2018 Jan;67:230-245. doi: 10.1016/j.bbi.2017.09.001. Epub 2017 Sep 7. PMID 28890155
- [Background] Haroon E, Welle JR, Woolwine BJ, Goldsmith DR, Baer W, Patel T, Felger JC, Miller AH. Associations among peripheral and central kynurenine pathway metabolites and inflammation in depression. Neuropsychopharmacology. 2020 May;45(6):998-1007. doi: 10.1038/s41386-020-0607-1. Epub 2020 Jan 15. PMID 31940661
- [Background] Hendry D, Campbell A, Smith A, Hopper L, Straker L, O'Sullivan P. Movement quantity and quality: How do they relate to pain and disability in dancers? PLoS One. 2022 May 19;17(5):e0268444. doi: 10.1371/journal.pone.0268444. eCollection 2022. PMID 35587918
- [Background] Huang WJ, Chen WW, Zhang X. Endocannabinoid system: Role in depression, reward and pain control (Review). Mol Med Rep. 2016 Oct;14(4):2899-903. doi: 10.3892/mmr.2016.5585. Epub 2016 Aug 1. PMID 27484193
- [Background] Lee Y, Jo J, Chung HY, Pothoulakis C, Im E. Endocannabinoids in the gastrointestinal tract. Am J Physiol Gastrointest Liver Physiol. 2016 Oct 1;311(4):G655-G666. doi: 10.1152/ajpgi.00294.2015. Epub 2016 Aug 18. PMID 27538961
- [Background] Lin TW, Kuo YM. Exercise benefits brain function: the monoamine connection. Brain Sci. 2013 Jan 11;3(1):39-53. doi: 10.3390/brainsci3010039. PMID 24961306
- [Background] Mackie K, Stella N. Cannabinoid receptors and endocannabinoids: evidence for new players. AAPS J. 2006 Apr 28;8(2):E298-306. doi: 10.1007/BF02854900. PMID 16796380
- [Background] Manca C, Boubertakh B, Leblanc N, Deschenes T, Lacroix S, Martin C, Houde A, Veilleux A, Flamand N, Muccioli GG, Raymond F, Cani PD, Di Marzo V, Silvestri C. Germ-free mice exhibit profound gut microbiota-dependent alterations of intestinal endocannabinoidome signaling. J Lipid Res. 2020 Jan;61(1):70-85. doi: 10.1194/jlr.RA119000424. Epub 2019 Nov 5. PMID 31690638
- [Background] McBride C, Bronner S. Injury characteristics in professional modern dancers: A 15-year analysis of work-related injury rates and patterns. J Sports Sci. 2022 Apr;40(7):821-837. doi: 10.1080/02640414.2021.2021030. Epub 2022 Jan 31. PMID 35100935
- [Background] Monda V, Villano I, Messina A, Valenzano A, Esposito T, Moscatelli F, Viggiano A, Cibelli G, Chieffi S, Monda M, Messina G. Exercise Modifies the Gut Microbiota with Positive Health Effects. Oxid Med Cell Longev. 2017;2017:3831972. doi: 10.1155/2017/3831972. Epub 2017 Mar 5. PMID 28357027
- [Background] Muccioli GG, Naslain D, Backhed F, Reigstad CS, Lambert DM, Delzenne NM, Cani PD. The endocannabinoid system links gut microbiota to adipogenesis. Mol Syst Biol. 2010 Jul;6:392. doi: 10.1038/msb.2010.46. PMID 20664638
- [Background] Nagy-Grocz G, Zador F, Dvoracsko S, Bohar Z, Benyhe S, Tomboly C, Pardutz A, Vecsei L. Interactions between the Kynurenine and the Endocannabinoid System with Special Emphasis on Migraine. Int J Mol Sci. 2017 Jul 30;18(8):1617. doi: 10.3390/ijms18081617. PMID 28758944
- [Background] Nunes AC, Mendes LA, Mota LA, Lima PO, Almeida GP. Training Load, Pain Intensity, and Functioning Can Explain Injuries in Dancers: A Classification and Regression Tree (CART) Analysis. Med Probl Perform Art. 2022 Jun;37(2):73-77. doi: 10.21091/mppa.2022.2012. PMID 35637559
- [Background] Purton T, Staskova L, Lane MM, Dawson SL, West M, Firth J, Clarke G, Cryan JF, Berk M, O'Neil A, Dean O, Hadi A, Honan C, Marx W. Prebiotic and probiotic supplementation and the tryptophan-kynurenine pathway: A systematic review and meta analysis. Neurosci Biobehav Rev. 2021 Apr;123:1-13. doi: 10.1016/j.neubiorev.2020.12.026. Epub 2021 Jan 19. PMID 33482244
- [Background] Rousseaux C, Thuru X, Gelot A, Barnich N, Neut C, Dubuquoy L, Dubuquoy C, Merour E, Geboes K, Chamaillard M, Ouwehand A, Leyer G, Carcano D, Colombel JF, Ardid D, Desreumaux P. Lactobacillus acidophilus modulates intestinal pain and induces opioid and cannabinoid receptors. Nat Med. 2007 Jan;13(1):35-7. doi: 10.1038/nm1521. Epub 2006 Dec 10. PMID 17159985
- [Background] Round JL, Mazmanian SK. The gut microbiota shapes intestinal immune responses during health and disease. Nat Rev Immunol. 2009 May;9(5):313-23. doi: 10.1038/nri2515. PMID 19343057
- [Background] Rudzki L, Ostrowska L, Pawlak D, Malus A, Pawlak K, Waszkiewicz N, Szulc A. Probiotic Lactobacillus Plantarum 299v decreases kynurenine concentration and improves cognitive functions in patients with major depression: A double-blind, randomized, placebo controlled study. Psychoneuroendocrinology. 2019 Feb;100:213-222. doi: 10.1016/j.psyneuen.2018.10.010. Epub 2018 Oct 16. PMID 30388595
- [Background] Russo F, Tolomeo F, Vandelli MA, Biagini G, Paris R, Fulvio F, Lagana A, Capriotti AL, Carbone L, Gigli G, Cannazza G, Citti C. Kynurenine and kynurenic acid: Two human neuromodulators found in Cannabis sativa L. J Pharm Biomed Anal. 2022 Mar 20;211:114636. doi: 10.1016/j.jpba.2022.114636. Epub 2022 Jan 31. PMID 35124451
- [Background] Saary P, Forslund K, Bork P, Hildebrand F. RTK: efficient rarefaction analysis of large datasets. Bioinformatics. 2017 Aug 15;33(16):2594-2595. doi: 10.1093/bioinformatics/btx206. PMID 28398468
- [Background] Shao BZ, Wei W, Ke P, Xu ZQ, Zhou JX, Liu C. Activating cannabinoid receptor 2 alleviates pathogenesis of experimental autoimmune encephalomyelitis via activation of autophagy and inhibiting NLRP3 inflammasome. CNS Neurosci Ther. 2014 Dec;20(12):1021-8. doi: 10.1111/cns.12349. PMID 25417929
- [Background] Shao BZ, Wang SL, Pan P, Yao J, Wu K, Li ZS, Bai Y, Linghu EQ. Targeting NLRP3 Inflammasome in Inflammatory Bowel Disease: Putting out the Fire of Inflammation. Inflammation. 2019 Aug;42(4):1147-1159. doi: 10.1007/s10753-019-01008-y. PMID 30937839
- [Background] Skonieczna-Zydecka K, Jakubczyk K, Maciejewska-Markiewicz D, Janda K, Kazmierczak-Siedlecka K, Kaczmarczyk M, Loniewski I, Marlicz W. Gut Biofactory-Neurocompetent Metabolites within the Gastrointestinal Tract. A Scoping Review. Nutrients. 2020 Nov 1;12(11):3369. doi: 10.3390/nu12113369. PMID 33139656
- [Background] Smid SD. Gastrointestinal endocannabinoid system: multifaceted roles in the healthy and inflamed intestine. Clin Exp Pharmacol Physiol. 2008 Nov;35(11):1383-7. doi: 10.1111/j.1440-1681.2008.05016.x. Epub 2008 Jul 29. PMID 18671715
- [Background] Yu W, Jin G, Zhang J, Wei W. Selective Activation of Cannabinoid Receptor 2 Attenuates Myocardial Infarction via Suppressing NLRP3 Inflammasome. Inflammation. 2019 Jun;42(3):904-914. doi: 10.1007/s10753-018-0945-x. PMID 30554372
- [Background] Wang X, He G, Peng Y, Zhong W, Wang Y, Zhang B. Sodium butyrate alleviates adipocyte inflammation by inhibiting NLRP3 pathway. Sci Rep. 2015 Aug 3;5:12676. doi: 10.1038/srep12676. PMID 26234821
- [Background] Wright KL, Duncan M, Sharkey KA. Cannabinoid CB2 receptors in the gastrointestinal tract: a regulatory system in states of inflammation. Br J Pharmacol. 2008 Jan;153(2):263-70. doi: 10.1038/sj.bjp.0707486. Epub 2007 Oct 1. PMID 17906675
- [Background] van Winden D, van Rijn RM, Savelsbergh GJP, Oudejans RRD, Stubbe JH. The Association Between Stress and Injury: A Prospective Cohort Study Among 186 First-Year Contemporary Dance Students. Front Psychol. 2021 Nov 5;12:770494. doi: 10.3389/fpsyg.2021.770494. eCollection 2021. PMID 34803856
- [Background] Sharkey KA, Wiley JW. The Role of the Endocannabinoid System in the Brain-Gut Axis. Gastroenterology. 2016 Aug;151(2):252-66. doi: 10.1053/j.gastro.2016.04.015. Epub 2016 Apr 29. PMID 27133395
- [Derived] Wiacek J, Podgorski T, Kusy K, Loniewski I, Skonieczna-Zydecka K, Karolkiewicz J. Evaluating the Impact of Probiotic Therapy on the Endocannabinoid System, Pain, Sleep and Fatigue: A Randomized, Double-Blind, Placebo-Controlled Trial in Dancers. Int J Mol Sci. 2024 May 21;25(11):5611. doi: 10.3390/ijms25115611. PMID 38891799